CLINICAL TRIAL: NCT06500182
Title: The Benefits of Hippotherapy for Patients With Parkinson's Disease of 75 Years of Age or More at Risk of Losing Their Independance.
Brief Title: The Benefits of Hippotherapy for Patients With Parkinson's Disease of 75 Years
Acronym: EQUIDIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A03105-34
Record Dates: First submitted 2021-05-20; First posted 2024-07-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hippotherapy sessions (Experimental): Patients will benefit from the hippotherapy sessions in additional to continuing to receive traditional care ,To evaluate any differences between the initial visit and the evaluation following 6 weeks in PDQ8 scores, which contain 8 items given a score between 0 (never) and 4 (always)
  Interventions: Other: hippotherapy sessions

INTERVENTIONS:
Other: hippotherapy sessions — Patients benefit from the hippotherapy sessions in additional to continuing to receive traditional care.

SUMMARY:
There is no cure for Parkinson's disease, resulting in an interest for research in this domain. Non pharmacological measures remain essential, specifically physical activity. Hippotherapy is a nonconventional method which uses the horse in addition to standard care. The goal being to improve or maintain the gains of the person through cognitive, sensorial and motor stimulation, with the aim of improving quality of life and maintaining independence. With this in mind, the researchers propose to evaluate quality of life as the main criterion, using the PDQ8 scale validated for this disease. The researchers hope results will lead to the coverage of the costs of non-conventional therapies such as hippotherapy by social security services.

DETAILED DESCRIPTION:
Parkinson's disease is a degenerative disorder with a prevalence of 2.50 patients per 1,000 people in 2015. Prevalence and incidence increase progressively with age up to the age of 80; more than half of patients are over 75.

There are two main types of Parkinson's disease in the elderly:

1. Parkinson's disease begins late, after the age of 75, and the disease may progress relatively slowly if there are no co-morbidities.
2. Or Parkinson's disease has been evolving for a long time, starting on average around the age of 55, and in this situation a number of difficulties arise depending on how long the disease has been present, the association of motor and non-motor fluctuations, the emergence of axonal signs and a decline in the severity of the disease, signs and a decline in cognitive function.

The therapeutic management of Parkinson's disease in the elderly must be assessed on a case-by-case basis. The efficacy/tolerance ratio of dopaminergic treatments must be taken into account.

In Alzheimer's disease (AD), it has been shown that aerobic exercise can delay cognitive decline. With this in mind, the researchers would like to propose a new and original approach using equitherapy in elderly Parkinson's patients.

The aim of this therapy will be to improve patients' quality of life, particularly in terms of well-being, maintain and encourage their autonomy and promote social interaction.

Equitherapy is an unconventional therapy which uses the horse as a complement to the treatment. For the EQUIDIA study, the researchers have suggested using the PDQ-8 score, validated for this condition, to evaluate quality of life as well as well-being and cognitive capacity for a group of Parkinson's patients over the age of 75 following 6 therapy sessions.Their Parkinson's diagnosis is to be confirmed through morphological and phase contrast MRI. The sessions will take place at the same interval of time following the administration of any dopaminergic medication. Progress will be recorded by the hippotherapy therapist using an evaluation developed by a horse-riding instructor. Sessions will be evaluated using inertia measurement devices to analyze quality of movement and the effect of specific activites with the horse.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years with PD according to Movement Disorders Society criteria (2015).
* Clinical diagnosis of Alzheimer's disease
* Has been on stable antiparkinsonian treatment for less than 3 months.
* Ability to understand the principle of the study as well as its risks.
* Written consent to participate in the trial.
* Have social insurance
* Agree to comply with all safety procedures during the study and its duration.
* Ability to understand and freely give consent
* Patient affiliated to social security or entitled beneficiary
* Autonomy preserved

Exclusion criteria :

* age <75 years
* refusal to sign consent
* MOCA <23
* Presence of major behavioural problems that do not allow MRI to be performed under optimal conditions
* Subjects unable to receive informed information, unable to participate in the study as a whole
* Subjects with a diagnosis of atypical parkinsonian syndrome (Lewy body disease, progressive supranuclear palsy, multisystem atrophy, cortico-basal degeneration, etc.).
* A classic contraindication to an MRI examination: claustrophobia, presence of incompatible foreign material,
* Subjects who have practised horse riding at a high level, animal phobias, wish to stop studying, etc.
* No affiliation to a social security scheme
* Antiparkinsonian treatment has not been stable for at least 3 months.
* People under protective supervision (guardianship, curatorship)
* People under family guardianship are also excluded, as are people for whom a mandate for future protection has been activated.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Assessing quality of life in Parkinson's disease by PDQ8 questionnaires | 06 weeks
  changes from baseline in PDQ8 scores, which contain 8 items given a score between 0 (never) and 4 (always) maximum control; range, 0 to 32.

SECONDARY OUTCOMES:
Assessing Parkinson's disease Motor disorders | 06 weeks
  Motor disorders assessed by Mbientlab devices .
Assessing Parkinson's disease severity of the non-motor symptoms | 06 weeks
  The severity of the non-motor symptoms of Parkinson's disease assessed by the score on the non-motor symptoms assesment scale for Parkinson's Disease. This is a 30-question questionnaire. For each question, a severity score ranging from 0 (none) to 3 (severe) and a frequency score ranging from 1 (rarely) to 4 (very frequent) are to be indicated.
Assessing Parkinson's disease Postural and walking disorders | 06 weeks
  Postural and walking disorders assessed by the Gait and Balance Scale (GABS) 33 (maximum control; range, 0 to 95). changes from baseline in severity motor signs of Parkinson's disease,assessed by the motor score of the MDS UPDRS scale.
MRI in diagnosis differential in Parkinson's disease | day 0
  The usefulness of flow MRI in diagnosis differential in Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga ATTIER, PHD, Principal Investigator — CH SAINT-QUENTIN
Locations (1):
- Centre Hospitalier de Saint-Quentin;, Saint-Quentin, Aisne, France

IPD SHARING:
Plan to Share IPD: No